CLINICAL TRIAL: NCT06196736
Title: An Open-label, Randomized Phase 3 Study to Evaluate 9MW2821 vs Investigator's Choice of Chemotherapy in Subjects With Locally Advanced or Metastatic Urothelial Cancer Who Have Previously Received PD-(L)1 Inhibitor and Platinum-containing Chemotherapy
Brief Title: A Study to Evaluate 9MW2821 Versus Chemotherapy in Subjects With Previously Treated Locally Advanced or Metastatic Urothelial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-2023-CP301
Record Dates: First submitted 2023-12-12; First posted 2024-01-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Advanced Urothelial Carcinoma
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW2821 (Experimental)
  Interventions: Drug: 9MW2821
- Investigator's Choice of Chemotherapy (Active Comparator)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: 9MW2821 — 1.25mg/kg of 9MW2821 by intravenous infusion on days 1, 8 and 15 of every 28-day cycle
  Arms: 9MW2821
Drug: Chemotherapy — 75mg/m^2 docetaxel by intravenous infusion or 175 mg/m^2 paclitaxel by intravenous infusion on day 1 of every 21-day cycle.
  Arms: Investigator's Choice of Chemotherapy

SUMMARY:
The purpose of this study was to compare the antitumor activity of 9MW2821 and chemotherapy in participants with locally advanced or metastatic urothelial cancer previously treated with PD-(L)1 inhibitor and platinum-containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to comprehend, sign, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form.
2. Male or female subjects aged 18 to 75 years (including 18 and 75 years).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed locally advanced or metastatic urothelial cancer, not amenable to resection with curative intent.
5. Subject must have received a platinum containing chemotherapy and PD-(L)1 inhibitor in the metastatic/locally advanced setting. If platinum and/or PD-(L)1 inhibitor was administered in the adjuvant/neoadjuvant setting subject must have progressed during treatment or within 12 months of completion.
6. Subject must have experienced radiographic progression during or after the last treatment regimen.
7. An archival tumor tissue sample or a fresh tissue sample should be provided.
8. Life expectancy of ≥ 12 weeks.
9. Subjects must have measurable disease according to RECIST (version 1.1).
10. Adequate organ functions.
11. Sexually active fertile subjects, and their partners, must agree to use methods of contraception during the study and at least 6 months after termination of study therapy.
12. Subjects are willing to follow study procedures.

Exclusion Criteria:

1. Chemotherapy or radiotherapy within 21 days prior to the first dose of study drug, traditional Chinese medicine with anticancer indication within 14 days prior to the first dose of study drug, use of any investigational drug or device within 28 days prior to the first dose of study drug, received treatment of nectin-4 targeted ADC, received treatment of ADC with MMAE payload, received prior chemotherapy with all available study therapies in the control arm, any strong CYP3A4 inducers/inhibitors within 14 days prior to the first dose of study drug.
2. Preexisting treatment related toxicity Grade ≥ 2 (except alopecia and grade 2 endocrine system toxicity with stable replacement therapy).
3. Major surgery within 28 days prior to first dose of study drug.
4. Hemoglobin A1C (HbA1c) ≥ 8%.
5. Preexisting peripheral neuropathy Grade ≥ 2.
6. Any live vaccines within 28 days before first dose of study drug or during the study.
7. Documented history of clinically significant cardiac or cerebrovascular diseases within 6 months prior to the first dose of study drug.
8. Other severe or uncontrolled disease, i.e. severe respiratory system disease, thromboembolic events, active bleeding or active infection.
9. Central nervous system metastases.
10. History of another malignancy within 3 years before the first dose of study drug. Subjects with cured malignancies are allowed.
11. History of autoimmune disease requiring systemic treatment within 2 years before the first dose of study drug.
12. Has ocular conditions that may increase the risk of corneal epithelium damage.
13. Known sensitivity to any of the ingredients of the investigational product; History of drug abuse or mental illness.
14. Uncontrolled tumor-related bone pain or spinal cord compression. Patients requiring pain medication must be on a stable regimen for at least 2 weeks before the first dose of study drug.
15. Pleural effusion, ascites or pericardial effusion with syptoms or needed drainage.
16. Condition or situation which may put the subject at significant risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival per Blinded Independent Central Review | Up to 3 years
  Time from the date of first randomization to the earliest date of documented disease progression per radiological evidence or death from any cause
Overall Survival | Up to 3 years
  Time from the date of randomization until the date of death from any cause

SECONDARY OUTCOMES:
Objective Response Rate per Blinded Independent Central Review and investigator | Up to 3 years
  The percentage of subjects who experience a best response of either CR or PR
Duration of Response per Blinded Independent Central Review and investigator | Up to 3 years
  Time from the date of the first complete response (CR) or partial response (PR) to the earliest date of disease progression or death from any cause
Time to response per Blinded Independent Central Review and investigator | Up to 3 years
  Time from the date of randomization to the date of confirmed CR or PR
Disease Control Rate per Blinded Independent Central Review and investigator | Up to 3 years
  Defined as the percentage of subjects who experience a best response of CR, PR or stable disease (SD)
Progression Free Survival per investigator | Up to 3 years
  Time from the date of first randomization to the earliest date of documented disease progression per radiological evidence or death from any cause
Incidence of adverse events | Up to 3 years
Incidence of Anti-Drug Antibody (ADA) | Up to 3 years
Mean change from baseline in the European Organisation for Research and Treatment of Cancer (EORTC) 30-item core quality-of-life questionnaire (QLQ-C30） | Up to 3 years
Mean change from baseline in EuroQOL 5-dimension 5-level Questionnaire [EQ-5D-5L] Visual Analog Scale (VAS) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang J, Liu R, Wang S, Feng Z, Yang H, Gao S, Li X, Yao X, Chen J, Gong Z, Li Y, Li X, Wang S, Hu C, Liu J, Zhang M, Yuan F, Shi B, Lou H, Zhao P, Qiu F, Guo H, Hu B, Xu D, Huang H, Zhang X, Feng M, Wang X, Li G, Liu D, Chen X, Wang P. Bulumtatug Fuvedotin (BFv, 9MW2821), a next-generation Nectin-4 targeting antibody-drug conjugate, in patients with advanced solid tumors: a first-in-human, open-label, multicenter, phase I/II study. Ann Oncol. 2025 Aug;36(8):934-943. doi: 10.1016/j.annonc.2025.04.009. Epub 2025 Apr 25. PMID 40288679